CLINICAL TRIAL: NCT05643144
Title: Enhancing Shared Decision-making to Prompt and Guide Individualized Care for People With Alzheimer's Disease and Diabetes
Brief Title: Enhancing Shared Decision-making to Guide Care for People With Dementia and Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, April Savoy, Assistant Professor, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13925; 1K01AG076971 (NIH)
Record Dates: First submitted 2022-11-11; First posted 2022-12-08 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-04

CONDITIONS: Diabetes; Alzheimer's Disease (Incl Subtypes); Dementia; Hypoglycemia
Keywords: Continuous glucose monitoring; Shared decision-making; Human factors; Primary care
MeSH Terms: conditions — Diabetes Mellitus; Alzheimer Disease; Dementia; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Patient-Caregiver Dyads (Experimental): Participants will wear a continuous glucose monitor
  Interventions: Device: Continuous Glucose Monitoring
- Patient-Caregiver Dyads & Clinicians (first iteration) (No Intervention): Participants will participate in the first iteration of the user-centered design process.
- Patient-Caregiver Dyads & Clinicians (second iteration) (No Intervention): Participants will participate in the second iteration of the user-centered design process.

INTERVENTIONS:
Device: Continuous Glucose Monitoring — CGM education and glucose data collection for 14 days with a device. Interviews with dyads to assess experience and awareness of hypoglycemic events.
  Arms: Patient-Caregiver Dyads

SUMMARY:
Aim 1: Characterize shared decision-making and unmet patient-caregiver dyads needs for patients with diabetes and Alzheimer's Disease and related dementias (ADRD) while using a continuous glucose monitoring (CGM) device.

Aim 2: Develop an interactive tool to enhance shared decision-making for diabetes management.

DETAILED DESCRIPTION:
Aim 1: Patient-caregiver dyads will participant in a semi-structured interview to establish a baseline. The dyad will receive standard diabetes educational materials along with a CGM training and instructions for device use. Patients will then wear the CGM device for 14 days. Three follow-up interviews will take place during the 14-day scanning period, as well as a debrief interview following the scanning period for assessment and technical support.

Aim 2: Patient-caregiver dyads and clinicians will participate in a user-centered design session to guide the design of interactive information displays to improve the interpretability of CGM data.

ELIGIBILITY:
Patient-Caregiver Dyad Inclusion Criteria (Aims 1 + 2):

* patient must have dual diagnosis of MCI or ADRD and diabetes (DM)
* patient must have active prescriptions for DM
* patient must have had at least one visit to an Eskenazi or IU Health primary care clinic within 12 months
* patient must be able to provide assent and have a legally authorized representative (LAR) consent on their behalf if patient lacks capacity to consent
* patient must have a caregiver aged 18 years or older who interacts daily, or almost daily, with the patient
* patient and caregiver must both speak English
* patient and caregiver must both reside in the community
* dyad must have internet access

Patient-Caregiver Dyad Exclusion Criteria (Aims 1 +2):

* patient has terminal illness
* use of an automated insulin delivery system
* patient is receiving dialysis
* patient is taking ascorbic acid during monitoring period
* patient has existing implanted medical devices
* patient has a bleeding disorder
* patient has a pre-existing arm skin lesions
* patient has an allergy to medical adhesive or isopropyl alcohol
* patient has plans for imaging or diathermy treatment during the study period

Clinician Participant Inclusion Criteria (Aim 2):

* primary care physicians
* nurses
* pharmacists
* nutritionists
* psychologists
* medical residents

Clinician Participant Exclusion Criteria (Aim 2):

* only treats patients younger than 65 years
* does not manage patients' DM

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2026-08-17 (Estimated); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Patient and Caregiver Unmet Needs (Aim 1) | 2 months
  Semi-structured Interviews: Baseline interview questions will be framed by validated psychometric measurements of hypoglycemia unawareness, fear of hypoglycemia, ADRD quality of life, and DM distress. Observation interviews will be conducted to elicit patients' and caregivers' perceptions about hypoglycemia and describe their specific risks (e.g., nutrition, resources, stress, finances). Debrief interviews will review CGM data with participants and ask clarifying questions to elicit descriptions of their overall experiences.
Level of Situation Awareness (Aim 2) | 1 day
  Contextual Inquiries: With and without examples of information displays present, we will invite participants questions related to identifying and reading glucose values (e.g., identify glycemic targets), and articulate perceived important information at specific decision points.

SECONDARY OUTCOMES:
Feasibility: Percentage of patients recruited (Aim 1) | 1 year
  Recruitment Percentage = Participant total/Eligible population total
Feasibility: Retention rate of participants (Aim 1) | 1 year
  Retention Rate = Completed participant total/Recruited participant total
Feasibility: CGM data completeness (Aim 1) | 2 months
  Count of total days CGM worn [CGM performs calculation]
Hypoglycemia: Percentage of time below range (Aim 1) | 2 months
  Percentage = glucose readings and time 54-69 mg/dL / total amount of readings and time monitored [CGM performs calculation]
Severe Hypoglycemia: Percentage of time below range (Aim 1) | 2 months
  Percentage = glucose readings and time <54 mg/dL / total amount of readings and time monitored [CGM performs calculation]
Percentage of time in range (Aim 1) | 2 months
  Percentage = glucose readings and time 70-180 mg/dL / total amount of readings and time monitored [CGM performs calculation]
Mean glucose (Aim 1) | 2 months
  Mean = sum of glucose readings / total amount of glucose readings [CGM performs calculation]
Glucose management indicator (Aim 1) | 2 months
  Estimated A1C automated calculation based on 14 days of CGM data [CGM performs calculation]
Glucose variability (Aim 1) | 2 months
  Oscillations in blood glucose levels: Measurement of fluctuations of glucose or other related parameters of glucose homoeostasis over a given interval of time (i.e., within a day, between days or longer term) [CGM performs calculation]

CONTACTS AND LOCATIONS:
Overall Officials: April Savoy, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Eskenazi Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No